CLINICAL TRIAL: NCT00643032
Title: Comparison of 2 Methods to Reduce Postoperative Pain in Children and a Comparison of 3 Methods of Preoperative Education Intervention to Reduce Anxiety in Children and Their Family
Brief Title: Preoperative Anxiety and Postoperative Pain in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Zvi Steiner, Hillel Yaffe Medical Center
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 50/2007
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Post-Operative Pain; Pre-Operative Anxiety
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator)
  Interventions: Procedure: Transcutaneous iliohypogastric
- II (Active Comparator)
  Interventions: Procedure: Perioperative administration near the nerve

INTERVENTIONS:
Procedure: Transcutaneous iliohypogastric
  Arms: I
Procedure: Perioperative administration near the nerve
  Arms: II

SUMMARY:
We wish to study which method of local injection of analgesic (before or during surgery) is the more effective method to reduce post-operative pain in children. In addition, we wish to study which pre-operative educational intervention is more effective in reducing anxiety in children and their family.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* ASA I - II
* Undergoing elective day surgery

Exclusion Criteria:

* Known coagulation dysfunction
* Sensitivity to analgesics

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel